CLINICAL TRIAL: NCT02744040
Title: Modulating the Impact of Critical Events in Early HIV Infection: Effect of ART Initiation and Alcohol Use
Acronym: MERLIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of California, San Francisco (Other); University of Washington (Other); Asociación Civil Impacta Salud y Educación, Peru (Other); Université de Montréal (Other); Seattle Children's Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ann C Duerr, Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA040532-01 (NIH); 8544 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1001540 (Other: Fred Hutch/University of Washington Cancer Consortium); R01DA040532-01 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-04-20 (Estimated); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: HIV Infection
Keywords: HIV reservoir; alcohol; ART
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early ART initiation (Other): Immediate ART initiation at the time of HIV diagnosis; daily dose of combination ART (one pill/day)
  Interventions: Drug: ART initiation at time of HIV diagnosis
- Deferred ART initiation (Other): ART initiation at 24 weeks after HIV diagnosis; daily dose of combination ART (one pill/day)
  Interventions: Drug: ART at 24 weeks

INTERVENTIONS:
Drug: ART initiation at time of HIV diagnosis — Immediate ART initiation
  Other Names: Early ART initiation
  Arms: Early ART initiation
Drug: ART at 24 weeks — ART initiation 24 weeks after enrollment
  Other Names: Deferred ART initiation
  Arms: Deferred ART initiation

SUMMARY:
The overall objective is to determine the influence of timing of ART initiation and alcohol consumption on HIV disease course. ART initiation immediately after HIV infection largely results in smaller HIV reservoir and lower HIV-associated systemic inflammation, which has been linked to non-AIDS morbidity and mortality. Immediate ART also reduces HIV-associated bacterial translocation and may prevent intestinal microbiome dysbiosis, that has been linked to increased systemic inflammation. Immediate intervention is not, however, generally feasible and more information is required about the consequences of starting ART at later time-points, but still early after acquisition. The study will be conducted in Lima, Peru, in a cohort of 180 MSM and transgender women (TW) with acute (Ab-, HIV RNA+) or recent (≤ 3 months) HIV infection. Alcohol use disorder (AUDIT score ≥8) is present in ~50% of HIV + participants in our cohort, four times higher than that seen among males in the general Peruvian population. Although the role of alcohol use in HIV pathogenesis and disease course remains unclear, some studies show a correlation with accelerated disease progression. The effects of alcohol resemble early post-infection changes in bacterial translocation and pro-inflammatory cytokines induced by HIV and their impact on HIV disease course before and after ART initiation remain unexplored.

Specific Aim 1: To determine the relative long-term benefits of immediate vs. early vs. delayed ART initiation at 24 weeks after diagnosis. The investigators will study outcomes after 2 and 4 years in MSM and TW diagnosed with acute or recent HIV infection.

Specific Aim 2: To determine the impact of alcohol use on the relative long-term benefits of immediate vs. early vs. delayed initiation of ART.

DETAILED DESCRIPTION:
Specific Aims: Recent studies suggest that very early initiation of ART (prior to seroconversion) does not prevent the establishment of HIV reservoirs, which eventually expand when ART is discontinued. Early ART initiation is, however, associated with preservation of CD4+ T cells and lower levels of total HIV DNA and cell-associated RNA as well as preservation of gut Th17 cells, thereby averting a major driver of HIV-related immune activation and limiting the size of the HIV reservoir. When, by contrast, ART is initiated in Fiebig III (FIII) or later, many HIV-associated changes have already occurred, including seeding of HIV reservoirs, damage to GI mucosa, and initiation of inflammatory cascades. Since ART initiation within weeks of HIV acquisition is not a viable public health strategy, it is important to more completely understand the relative long-term benefits of initiating ART at very early times after infection (FI-II) as opposed to after a short (during FIII-V) or longer delay (at 24 weeks). Since the possibility that high-level alcohol use can mitigate the benefits of early ART is emerging as a potentially important public health issue, the investigators will evaluate the impact of time of ART initiation as well as alcohol use on HIV pathogenesis in Peruvian men who have sex with men (MSM) and TW, in whom high-level alcohol use is common. They will study outcomes after 2 and 4 years in MSM and TW diagnosed with acute (Ab-, HIV RNA+) or recent (≤3 months) HIV infection. Three groups based on time since estimated date of detectible HIV infection (EDDI) to ART initiation will be studied: a) EDDI-to-ART: ≤ 30 days b) EDDI-to-ART: 31-90 days and c) EDDI-to-ART: >90 days

The overarching hypotheses are: 1. Initiation of ART soon after HIV infection will dampen perturbations of GI microbiota, reduce HIV-induced inflammatory changes, and decrease seeding of the reservoir. Initiation of ART within 30 days will have the greatest benefit. 2. Irrespective of the time of ART initiation, alcohol use will compound the negative effects of HIV.

SPECIFIC AIM 1) To determine the relative long-term benefits of immediate vs. early vs. delayed initiation of ART. Initiation of ART within 30 days of infection, while theoretically appealing, is infeasible in clinical practice because antibody-based tests, used almost world-wide, are unable to diagnose very early infection. Six months of ART initiated shortly after seroconversion can improve many immune parameters, although not to the near normal level seen when ART is initiated earlier.. Longer-term follow-up of seropositive participants who started ART ~2-8 months after HIV acquisition compared to those initiating ART within 30 days is needed to see whether markers of inflammation and residual viral load might continue to improve after 6 months, decreasing the difference between the groups. Methods: the investigators will evaluate the 3 groups using specimens from equivalent times after ART initiation for a total of 4 years of ART, comparing viral load, CD4 counts, time to reach undetectable VL, the GI microbiota, and inflammatory markers. Specimens from uninfected and chronically infected subjects are available as controls for some outcomes. They will model the size and persistence of the viral reservoir across all ART-compliant study subjects, measuring total HIV DNA, integrated HIV DNA and multi-spliced HIV RNA via TILDA (Tat/Rev Induced Limiting Dilution Assay) assay. In a subset of individuals from each group, the proviral integration sites will be defined at ART initiation and after 2 and 4 years to assess the maintenance of the reservoir by proliferating CD4 cells.

SPECIFIC AIM 2) To determine the impact of high-level alcohol use on the relative long-term benefits of immediate vs. early vs. delayed ART initiation. High-level alcohol use results in changes in the GI microbiome, increasing dysbiosis and gut permeability, and these changes are associated with up-regulation of inflammatory pathways.. Dysbiosis is present in many HIV-infected patients. Methods: Investigators will compare outcomes between subjects by their reported alcohol use or by assessing alcohol use blood biomarkers (Phosphatidylethanol; PEth) at specified timepoints.. Finally, among ART-adherent subjects with persistent viral suppression, the investigators will assess inflammatory markers and HIV reservoirs in those with and without high-level alcohol use at 2 and 4 years after ART initiation.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men or transgender women HIV-infected with prior participation in SABES study in Lima Peru OR Established HIV infection OR HIV uninfected

Exclusion Criteria:

* counter-indication for use of study antiretroviral drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Duerr, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Asociación Civil Impacta Salud y Educación, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Massanella M, Ignacio RAB, Lama JR, Pagliuzza A, Dasgupta S, Alfaro R, Rios J, Ganoza C, Pinto-Santini D, Gilada T, Duerr A, Chomont N. Long-term effects of early antiretroviral initiation on HIV reservoir markers: a longitudinal analysis of the MERLIN clinical study. Lancet Microbe. 2021 May;2(5):e198-e209. doi: 10.1016/s2666-5247(21)00010-0. Epub 2021 Mar 23. PMID 34841369

RESULTS

PARTICIPANT FLOW:
Groups:
- EDDI-to-ART <= 30 Days: Participants who started ART within 30 days from the estimated date of infection
- EDDI-to-ART 31-90 Days: Participants who started ART between 31 and 90 days from the estimated date of infection
- EDDI-to-ART >90 Days: Participants who started ART more than 90 days from the estimated date of infection
Period: Overall Study
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Started | 28 | 51 | 72
Completed | 22 | 40 | 50
Not Completed | 6 | 11 | 22
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Physician Decision | 0 | 8 | 13
Not completed — Lost to Follow-up | 3 | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days | Total
Number analyzed (Participants) | 28 | 51 | 72 | 151
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [24 to 30] | 26 [22 to 31] | 24 [21 to 30] | 25 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 28 | 51 | 72 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 51 | 72 | 151
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 28 | 51 | 72 | 151
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Peru | 28 | 51 | 72 | 151
HIV Viral Load [Median (Inter-Quartile Range); unit: Log10(Copies/mL)] | 6.6 [5.8 to 7.0] | 5.4 [4.8 to 6.3] | 5.8 [5.0 to 6.6] | 5.8 [5.0 to 6.7]
CD4 count [Median (Inter-Quartile Range); unit: Cells/mm3] | 521 [300 to 595] | 428 [206 to 554] | 421 [299 to 567] | 442 [282 to 572]

OUTCOME MEASURES:

1. Primary Outcome: Baseline HIV DNA Reservoir: Total HIV DNA
Description: Total HIV DNA reservoir at baseline (ART Initiation) Baseline total HIV DNA was measured in CD4+ T cells isolated from PBMC collected at the ART Initiation visit. Total DNA was quantitated using polymerase chain reaction (PCR) with primers within HIV (5'-LTR and gag).
Time Frame: Baseline
Population: The number of participants in the analysis of individual outcomes at some timepoints differs from the total number of participants shown in the participant flow due to lack of specimen availability and missed visits for some participants. In addition, some analyses were only conducted in selected participants (for example, restriction to participants with baseline specimens).
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 9 | 14 | 19
Log10 HIV DNA copies/10^6 CD4 T cells | 3.83 [3.45 to 3.99] | 3.67 [3.24 to 4.13] | 3.40 [2.81 to 3.72]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; Total HIV DNA at the time of ART initiation in each of the three EDDI groups; Test type: Other; p = 0.048, Mixed Effects Models — Multiple hypothesis testing was performed using Tukey's Honest Significant Difference (HSD) procedure

2. Primary Outcome: Two Phase Decay of HIV DNA Reservoir: Total HIV DNA
Description: Decay of total HIV DNA was assessed in CD4+ T cells isolated from PBMC collected at 1, 2, 4, 8, 16, 24, 96 and 192 weeks (as available) from ART initiation (which occurred prior to enrollment into MERLIN). Total DNA was quantitated using polymerase chain reaction (PCR) with primers within HIV (5'-LTR and gag). The longitudinal decay in total HIV DNA was analyzed by use of a mixed-effects model from the time of ART initiation up to 192 weeks.
Time Frame: 4 years from ART initiation
Population: The number of participants in the analysis of individual outcomes at some timepoints differs from the total number of participants shown in the participant flow due to lack of specimen availability and missed visits for some participants. In addition, some analyses were only conducted in selected participants (for example, restriction to participants with baseline specimens or participants with continuous viral load suppression after ART initiation).
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells/WK
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 9 | 14 | 19
Log10 HIV DNA copies/10^6 CD4 T cells/WK
  Slope 1 | -0.145 [-0.164 to -0.126] | -0.058 [-0.067 to -0.050] | -0.018 [-0.021 to -0.015]
  Slope 2 | -0.006 [-0.007 to -0.005] | -0.004 [-0.005 to -0.003] | -0.001 [-0.002 to 0.001]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; The decay in total HIV DNA was modeled from the time of ART initiation in each of the three EDDI groups until the end of follow-up. The decay was analyzed on the log10 scale with a mixed-effects model to account for correlation between measurements from the same individual. We used a piecewise linear function to model the decay, where the number of linear segments was fixed at 2 (two-phase segmentation model) for Total HIV DNA; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-wise comparison of Slope 1
Statistical Analysis 2: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-wise comparison of Slope 1
Statistical Analysis 3: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-wise comparison of Slope 1
Statistical Analysis 4: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 5: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 6: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 2, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2

3. Primary Outcome: Baseline HIV DNA Reservoir: Integrated HIV DNA
Description: Baseline integrated HIV DNA was measured in CD4+ T cells isolated from PBMC collected at the ART Initiation visit. Integrated DNA was quantitated using polymerase chain reaction (PCR) with primers within HIV (3'-LTR) and host DNA (alu).
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 9 | 14 | 19
Log10 HIV DNA copies/10^6 CD4 T cells | 2.87 [2.80 to 3.26] | 2.76 [2.24 to 3.20] | 2.55 [2.23 to 2.97]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; Integrated HIV DNA at the time of ART initiation in each of the three EDDI groups; Test type: Other; p > 0.05, Mixed Effects Models — Multiple hypothesis testing was performed using Tukey's HSD procedure

4. Primary Outcome: Two Phase Decay of HIV DNA Reservoir: Integrated HIV DNA
Description: Decay of integrated HIV DNA was assessed in CD4+ T cells isolated from PBMC collected at 1, 2, 4, 8, 16, 24, 96 and 192 weeks (as available) from ART initiation (which occurred prior to enrollment into MERLIN).. Integrated DNA was quantitated using polymerase chain reaction (PCR) with primers within HIV (3'-LTR) and host DNA (alu). The longitudinal decay in integrated HIV DNA was analyzed by use of a mixed-effects model from the time of ART initiation up to 192 weeks.
Time Frame: 4 years from ART initiation
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells/WK
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 9 | 14 | 19
Log10 HIV DNA copies/10^6 CD4 T cells/WK
  Slope 1 | -0.149 [-0.174 to -0.124] | -0.049 [-0.060 to -0.038] | -0.014 [-0.019 to -0.010]
  Slope 2 | -0.002 [-0.003 to -0.001] | -0.001 [-0.002 to 0.000] | -0.001 [-0.002 to 0.000]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; The decay in integrated HIV DNA was modeled from the time of ART initiation in each of the three EDDI groups until the end of follow-up. The decay was analyzed on the log10 scale with a mixed-effects model to account for correlation between measurements from the same individual. We used a piecewise linear function to model the decay, where the number of linear segments was fixed at 2 (two-phase segmentation model) for integrated HIV DNA; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 2: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 4, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 3: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 4, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 4: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; [analysis description as in outcome 4, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 5: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 4, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 6: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 4, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2

5. Primary Outcome: Baseline HIV DNA Reservoir: TILDA Stimulation
Description: Baseline HIV DNA by TILDA stimulation was measured in CD4+ T cells isolated from PBMC collected at the ART Initiation visit. The inducible HIV reservoir (TILDA stimulation) was quantitated using a tat/rev induced limiting dilution assay (TILDA). Cells with inducible HIV proviruses were assessed by quantifying the frequency of CD4+ cells producing multiply-spliced HIV RNA after in-vitro stimulation.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 5 | 10 | 17
Log10 HIV DNA copies/10^6 CD4 T cells | 2.94 [1.60 to 3.14] | 2.02 [1.80 to 2.56] | 1.66 [1.21 to 2.14]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; TILDA stimulation reservoir measure at the time of ART initiation in each of the three EDDI groups; Test type: Other; p = 0.057, Mixed Effects Models — Multiple hypothesis testing was performed using Tukey's HSD procedure

6. Primary Outcome: Two Phase Decay of HIV DNA Reservoir: TILDA Stimulation
Description: Decay of inducible HIV DNA proviruses (TILDA stimulation) was assessed in CD4+ T cells isolated from PBMC collected at 1, 2, 4, 8, 16, 24, 96 and 192 weeks (as available) from ART initiation (which occurred prior to enrollment into MERLIN). The inducible HIV reservoir (TILDS stimulation) was quantitated using a tat/rev induced limiting dilution assay (TILDA). Cells with inducible HIV proviruses were assessed by quantifying the frequency of CD4+ cells producing multiply-spliced HIV RNA after in-vitro stimulation. The longitudinal decay in the inducible HIV DNA reservoir was analyzed by use of a mixed-effects model from the time of ART initiation up to 192 weeks.
Time Frame: 4 years from ART initiation
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Log10 HIV DNA copies/10^6 CD4 T cells/WK
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 5 | 10 | 17
Log10 HIV DNA copies/10^6 CD4 T cells/WK
  Slope 1 | -0.266 [-0.311 to -0.221] | -0.170 [-0.204 to -0.136] | -0.143 [-0.170 to -0.115]
  Slope 2 | -0.002 [-0.003 to 0.000] | -0.001 [-0.002 to 0.001] | 0.001 [0.000 to 0.002]
Statistical Analysis 1: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; The decay in TILDA stimulation was modeled from the time of ART initiation in each of the three EDDI groups until the end of follow-up. The decay was analyzed on the log10 scale with a mixed-effects model to account for correlation between measurements from the same individual. We used a piecewise linear function to model the decay, where the number of linear segments was fixed at 2 (two-phase segmentation model) for TILDA Stimulation; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p = 0.010, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 2: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 6, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p < 0.0001, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 3: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 6, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 1
Statistical Analysis 4: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART 31-90 Days; [analysis description as in outcome 6, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 5: Comparison: EDDI-to-ART <= 30 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 6, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p = 0.052, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2
Statistical Analysis 6: Comparison: EDDI-to-ART 31-90 Days vs EDDI-to-ART >90 Days; [analysis description as in outcome 6, analysis 1]; Test type: Other — Tukey's Honest Significant Difference (HSD) test; p > 0.05, Tukey's Honest Significant Difference (H — Pair-Wise comparison of Slope 2

7. Primary Outcome: HIV DNA Integration Sites
Description: HIV DNA integration sites were measured for up to 4 years after initiation of ART (which occurred prior to enrollment in MERLIN). HIV DNA integration was assessed using CD4+ T cells isolated from PBMC at enrollment, ART initiation and 24, 96 and 192 weeks after ART initiation. HIV integration into the STAT5 and BACH2 genes was measured by assessing hybrid transcript structure (HIV LTR to BACH2 or STAT5 exon); hybrid transcript structure was confirmed by sequencing.
Time Frame: 4 years from ART initiation
Population: Specimen collection has been completed but the analysis could not be completed due to unforeseen circumstances.
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: GI Microbiome
Description: The GI microbiome will be assessed using 16S rRNA-based phylogenetic characterization of microbiome composition using stool specimens obtained before and after ART initiation.
Time Frame: 4 years from ART initiation
Population: Specimen collection has been completed but the analysis could not be completed due to unforeseen circumstances.
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Levels of Inflammatory Markers
Description: Levels of inflammatory biomarkers measured in plasma by Meso Scale Discovery (MSD) and ELISA assays prior to infection and after viral load suppression.
Time Frame: 4 years from ART initiation
Population: Specimen collection has been completed but the analysis could not be completed due to unforeseen circumstances.
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Impact of Alcohol Use
Description: High level alcohol use will be measured using self report (AUDIT Score and Quick Drinking Survey) and a blood biomarker (PEth). Alcohol use level will be included in multivariate analysis of GI Microbiome composition as well as a covariate in other analyses.
Time Frame: 4 years from ART initiation
Population: Specimen collection has been completed but the analysis could not be completed due to unforeseen circumstances.
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 0 | 0 | 0

11. Primary Outcome: HIV RNA Viral Load
Description: HIV viral load was measured in plasma at multiple timepoints beginning with the first visit after HIV diagnosis (which occurred prior to enrollment in MERLIN), using standard commercial viral load kits with a cut-off of 40 HIV RNA copies/mL. The log10 of HIV RNA copies/mL is reported. A value of 1.6 or less represent an undetectable log10 viral load (log10 <40 copies/mL).
Time Frame: 4 years from ART initiation
Measure: Median (Inter-Quartile Range); unit: Log10 HIV RNA copies/mL
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 28 | 51 | 72
Log10 HIV RNA copies/mL
  At ART Initiation | 6.63 [6.06 to 7] | 5.42 [4.82 to 6.385] | 4.96 [4.60 to 5.53]
  One year on ART | 1.6 [0 to 1.6] | 1.6 [0 to 1.6] | 1.6 [0 to 1.6]
  Two years on ART | 1.6 [0 to 1.6] | 1.6 [0 to 1.6] | 1.6 [0 to 1.6]
  Three years on ART | 1.6 [0 to 1.6] | 1.6 [0 to 1.6] | 1.6 [0 to 1.6]
  Four years on ART | 1.6 [0 to 1.6] | 1.6 [0 to 1.6] | 1.6 [0 to 1.6]

12. Primary Outcome: CD4 Count
Description: CD4 counts were measured by flow cytometry at multiple timepoints in all participants.
Time Frame: 4 years from ART initiation
Measure: Median (Inter-Quartile Range); unit: Cells/mm^3
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 28 | 51 | 72
Cells/mm^3
  At ART Initiation | 656 [564 to 724] | 609 [377 to 754] | 552 [452 to 700]
  One year on ART | 622 [525 to 770] | 584 [473 to 738] | 635 [502 to 795]
  Two years on ART | 653 [599 to 919] | 595 [396 to 781] | 696 [550 to 902]
  Three years on ART | 675 [592 to 846] | 703 [493 to 820] | 706 [586 to 874]
  Four years on ART | 707 [610 to 985] | 643 [516 to 790] | 690 [535 to 850]

13. Primary Outcome: Time to Undetectable HIV Viral Load
Description: Number of days between ART start and Undetectable Viral Load (<40 copies/mL)
Time Frame: 4 years from ART initiation
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
Number analyzed (Participants) | 26 | 47 | 63
Days | 163.5 [84 to 171.25] | 110 [84 to 169] | 154 [84 to 168]

ADVERSE EVENTS:
Time Frame: Up to 3 years and 3 months
Arm/Group | EDDI-to-ART <= 30 Days | EDDI-to-ART 31-90 Days | EDDI-to-ART >90 Days
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/51 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/51 | 1/72
Other Adverse Events (participants affected / at risk) | 14/28 | 26/51 | 46/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDDI-to-ART <= 30 Days (N=28) | EDDI-to-ART 31-90 Days (N=51) | EDDI-to-ART >90 Days (N=72)
rectal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EDDI-to-ART <= 30 Days (N=28) | EDDI-to-ART 31-90 Days (N=51) | EDDI-to-ART >90 Days (N=72)
Hemorrhoids (Gastrointestinal disorders) | 5 | 5 | 9
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 10
Pharyngitis (Infections and infestations) | 2 | 2 | 5
SARS-Cov-2 Infection (COVID-19 Disease) (Infections and infestations) | 1 | 3 | 2
Syphilis (Infections and infestations) | 6 | 14 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02744040/Prot_000.pdf